CLINICAL TRIAL: NCT01479465
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GS-6624 Combined With FOLFIRI as Second Line Treatment for Metastatic KRAS Mutant Colorectal Adenocarcinoma That Has Progressed Following a First Line Oxaliplatin- and Fluoropyrimidine-Containing Regimen
Brief Title: Efficacy and Safety of Simtuzumab (SIM) With FOLFIRI as Second Line Treatment in Colorectal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-295-0203; 2011-003754-61 (EudraCT Number)
Record Dates: First submitted 2011-11-09; First posted 2011-11-24 (Estimated); Results first posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
Keywords: GSI; Gilead; Gilead Sciences; GS-6624; Colorectal Cancer; KRAS; Oncology; monoclonal antibody
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms | interventions — simtuzumab; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FOLFIRI + SIM 700 mg (Part A) (Experimental): Participants will receive SIM 700 mg via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Biological: Simtuzumab; Drug: Leucovorin; Drug: Irinotecan; Drug: Fluorouracil
- FOLFIRI + SIM 200 mg (Part B) (Experimental): Participants will receive SIM 200 mg via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Biological: Simtuzumab; Drug: Leucovorin; Drug: Irinotecan; Drug: Fluorouracil
- FOLFIRI + SIM 700 mg (Part B) (Experimental): Participants will receive SIM 700 mg via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Biological: Simtuzumab; Drug: Leucovorin; Drug: Irinotecan; Drug: Fluorouracil
- FOLFIRI + Placebo (Part B) (Experimental): Participants will receive placebo to match SIM via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Placebo to match SIM; Drug: Leucovorin; Drug: Irinotecan; Drug: Fluorouracil

INTERVENTIONS:
Biological: Simtuzumab — SIM administered via intravenous infusion over 30 minutes
  Other Names: SIM; GS-6624
  Arms: FOLFIRI + SIM 200 mg (Part B); FOLFIRI + SIM 700 mg (Part A); FOLFIRI + SIM 700 mg (Part B)
Drug: Placebo to match SIM — Placebo to match SIM administered via intravenous infusion over 30 minutes
  Arms: FOLFIRI + Placebo (Part B)
Drug: Leucovorin — l-Leucovorin 200 mg/m^2 or dl-leucovorin 400 mg/m^2 administered via intravenous infusion over 2 hours
  Other Names: Folinic acid
Drug: Irinotecan — Irinotecan 180 mg/m^2 administered via intravenous infusion over 90 minutes
Drug: Fluorouracil — Fluorouracil 400 mg/m^2 administered via intravenous bolus and 2400 mg/m^2 via intravenous infusion over 46 hours

SUMMARY:
The primary objective of this study is to compare the additive efficacy of SIM versus placebo in combination with leucovorin (folinic acid), irinotecan, and fluorouracil (FOLFIRI) as measured by improvement in progression-free survival (PFS) in participants with metastatic KRAS mutant colorectal adenocarcinoma who have progressed following a first-line oxaliplatin- and fluoropyrimidine-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal carcinoma with KRAS mutation
* Received first line therapy and discontinued part or all of first line therapy
* Estimated life expectancy > 3 months
* Stage IV disease
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* Adequate hepatic and hematologic function
* No major operations within 4 weeks prior to treatment start

Exclusion Criteria:

* More than 1 prior chemotherapy regimen for Stage 4 colorectal cancer
* Experimental medical treatment within 30 days prior to study entry
* Known or suspected cerebral metastases
* History or presence of any form of cancer, other that colorectal cancer, within the 3 years prior to enrollment
* Known dihydropyrimidine dehydrogenase-deficiency (special screening not required)
* Subjects with angina pectoris, poorly controlled ventricular arrhythmias (does not include asymptomatic, occasional premature ventricular contractions), history of clinically significant coronary heart disease or cardiomyopathy, or electrocardiogram (ECG) abnormalities consistent with ischemia
* Uncontrolled hypertension (seated systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg) at screening
* Clinically active liver disease, including active hepatitis (any etiology) or cirrhosis
* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, hormonal therapy) within 21 days prior to randomization
* Prior irinotecan therapy for metastatic disease is not permitted
* Systemic fungal, bacterial, viral, or other infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zung Thai, MD, Study Director — Gilead Sciences
Locations (109):
- United States (56):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Providence Saint Joseph Medical Center-Disney Family Cancer Center, Burbank, California
  - Wilshire Oncology Medical Group, Inc., Corona, California
  - Saint Jude Heritage Healthcare, Fullerton, California
  - University of California San Diego Medical Center, La Jolla, California
  - Pacific Shores Medical Group, Long Beach, California
  - Comprehensive Hematology Oncology Centers, Inc., Los Angeles, California
  - TORI Network (Translational Oncology Research Intl), Los Angeles, California
  - UCLA Community Oncology Practice, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Wilshire Oncology Medical Group, Inc., Pomona, California
  - Cancer Care Associates Medical Group, Redondo Beach, California
  - Pacific Shores Medical Group, Redondo Beach, California
  - Sharp Health Care, San Diego, California
  - San Jose Medical Group, San Jose, California
  - Central Coast Medical Oncology Corp, Santa Maria, California
  - Yale University Smilow Cancer Hospital, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Gainesville, Florida
  - MD Anderson Cancer Center, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Peachtree Hematology Oncology Consultants, PC, Atlanta, Georgia
  - Suburban Hematology Oncology Associates, PC, Lawrenceville, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Hematology and Oncology Associates at BridgePoint, Tupelo, Mississippi
  - Saint Joseph Oncology, Inc., Saint Joseph, Missouri
  - Montana Cancer Institute, Missoula, Montana
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York University Clinical Cancer Center, New York, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Oncology Hematology Care, Inc., Wilmington, Ohio
  - Kaiser Permanente Northwest Region Oncology Hematology, Portland, Oregon
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Center for Cancer and Blood Disorders, PC, Fort Worth, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Scott & White Memorial, Temple, Texas
  - The Center for Cancer and Blood Disorders, Weatherford, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Intermountain Healthcare, St. George, Utah
  - Virginal Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Institute, Midlothian, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- France (8):
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Auvergne
  - Centre Eugène Marquis, Rennes, Brittany Region
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Dept. de Cancerologie Digestive et Urologique, Lille
  - Centre Hospitalier Régional Universitaire Hôpital Saint Eloi, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Paoli Calmettes Centre Régional de Lutte Contre le Cancer, Rennes
  - Hôpital Trousseau - Service de Gastroenterologie, Tours
- Germany (13):
  - Universitätsklinikums Mannheim, Mannheim, Baden-Wuerttenberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Ludwig-Maximilians-Universität München Klinikum Großhadern, München, Bavaria
  - Klinikum Region Hannover GmbH, Krankenhaus Siloah, Hanover, Lower Saxony
  - Universitätsklinikum Rostock, Rostock, Mecklenburg-Vorpommern
  - Medizinische Universitätsklinik Bochum, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Krankenanstalt Mutterhaus der Borromäerinnen e.V., Trier, Rhineland-Palatinate
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum der Friedrich-Schiller-Universität Jena, Jena, Thuringia
  - Städtisches Klinikum Frankfurt-Höchst, Frankfurt
  - Katholisches Marienkrankenhaus gGmbH, Hamburg
  - University Magdeburg, Magdeburg
- Italy (6):
  - Ospedale Unico Versilia, Lido di Camaiore, Lucca
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Monza E Brianza
  - Arcispedale Santa Maria Nuova IRCCS, Reggio Emilia, Reggio Nella Emilia
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Niguarda Cà Granda, Milan
  - Ospedale Civile SS Annunziata ASL 1, Sassari
- Poland (6):
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Spólka z o. o., Krakow, Lesser Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Olsztynski Osrodek Onkologiczny "Kopernik" sp. z o. o., Olsztyn, Warmian-Masurian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Centrum Onkologii - Instytut im Marii Sklodowskiej-Curie, Warsaw
- Russia (9):
  - State Institution of Healthcare "Arkhangelsk Regional Clinical Oncology Dispensary", Arkhangelsk
  - Republican Clinical Oncologic Dispensary of Ministry of health of Republic Tatarstan, Kazan'
  - Kursk Regional Oncologic Dispensary, Kursk
  - Cancer Research Center n.a. Blokhin, Chemotherapy Dept., Moscow
  - Non-State Institution of healthcare "Central Clinical Hospital #1 OAO RZD", Moscow
  - State Institution "Blokhin Cancer Research Centre RAMS", Moscow
  - Nizhny Novgorod City Oncology Dispensary, Nizhny Novgorod
  - State Healthcare Institution of Omsk Region "Clinical Oncologic Dispensary", Omsk
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg
- Spain (11):
  - Centro Oncológico Regional de Galicia, A Coruña, La Coruna
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Hospital de Madrid Norte-San Chinarro, Madrid
  - Hospital Universitario La Paz, Madrid
  - Instituto de Investigación Sanitaria, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Hecht JR, Benson AB 3rd, Vyushkov D, Yang Y, Bendell J, Verma U. A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Simtuzumab in Combination with FOLFIRI for the Second-Line Treatment of Metastatic KRAS Mutant Colorectal Adenocarcinoma. Oncologist. 2017 Mar;22(3):243-e23. doi: 10.1634/theoncologist.2016-0479. Epub 2017 Feb 28. PMID 28246207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Russia, and Europe. The first participant was screened on 15 December 2011. The last study visit occurred on 27 February 2015.
Pre-assignment Details: 358 participants were screened.
Groups:
- FOLFIRI + SIM 700 mg (Part A): Participants received simtuzumab (SIM) 700 mg via intravenous infusion followed by leucovorin (folinic acid), irinotecan, and fluorouracil (FOLFIRI; l-leucovorin 200 mg/m^2 or dl-leucovorin 400 mg/m^2 administered via intravenous infusion over 2 hours and irinotecan 180 mg/m^2 administered via intravenous infusion over 90 minutes, followed by fluorouracil 400 mg/m^2 administered via intravenous bolus and 2400 mg/m^2 via intravenous infusion over 46 hours) on Days 1 and 15 of each 28-day treatment cycles for approximately 10 months.
- FOLFIRI + Placebo (Part B): Participants received placebo to match SIM via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycles for approximately 27 months.
- FOLFIRI + SIM 200 mg (Part B): Participants received SIM 200 mg via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycles for approximately 21 months.
- FOLFIRI + SIM 700 mg (Part B): Participants received SIM 700 mg via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycles for approximately 19 months.
Period: Overall Study
Arm/Group | FOLFIRI + SIM 700 mg (Part A) | FOLFIRI + Placebo (Part B) | FOLFIRI + SIM 200 mg (Part B) | FOLFIRI + SIM 700 mg (Part B)
Started | 11 | 84 | 86 | 85
Completed | 0 | 0 | 0 | 0
Not Completed | 11 | 84 | 86 | 85
Not completed — Disease Progression | 9 | 61 | 65 | 70
Not completed — Study Discontinued by Sponsor | 0 | 7 | 5 | 3
Not completed — Adverse Event | 0 | 3 | 6 | 4
Not completed — Investigator Discretion | 1 | 4 | 2 | 4
Not completed — Subject Request | 1 | 3 | 4 | 2
Not completed — Subject Withdrew Consent | 0 | 5 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were analyzed.
Groups:
- FOLFIRI + SIM 700 mg (Part A): Participants received SIM 700 mg via intravenous infusion followed by FOLFIRI via intravenous infusion on Days 1 and 15 of each 28-day treatment cycles for approximately 10 months.
- Total: Total of all reporting groups
Arm/Group | FOLFIRI + SIM 700 mg (Part A) | FOLFIRI + Placebo (Part B) | FOLFIRI + SIM 200 mg (Part B) | FOLFIRI + SIM 700 mg (Part B) | Total
Number analyzed (Participants) | 11 | 84 | 86 | 85 | 266
Age, Customized [Count of Participants; unit: Participants] — Full Analysis Set included participants who were randomized and received at least 1 dose of study drug. Population: Participants in Full Analysis Set were analyzed.
  Participants
    number analyzed (Participants) | 11 | 80 | 85 | 84 | 260
    Between 18 and 65 years | 7 | 57 | 49 | 56 | 169
    ≥ 65 years | 4 | 23 | 36 | 28 | 91
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants in Full Analysis Set were analyzed.
  Participants
    number analyzed (Participants) | 11 | 80 | 85 | 84 | 260
    Female | 6 | 41 | 32 | 48 | 127
    Male | 5 | 39 | 53 | 36 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in Full Analysis Set were analyzed.
  Participants
    Race: number analyzed (Participants) | 11 | 80 | 85 | 84 | 260
    Race: White | 8 | 67 | 74 | 71 | 220
    Race: Black or African American | 2 | 8 | 5 | 7 | 22
    Race: Asian | 1 | 1 | 5 | 1 | 8
    Race: Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1 | 2
    Race: Not Permitted | 0 | 3 | 1 | 3 | 7
    Race: Missing | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants in Full Analysis Set were analyzed.
  Participants
    Ethnicity: number analyzed (Participants) | 11 | 80 | 85 | 84 | 260
    Ethnicity: Non-Hispanic/Latino | 8 | 70 | 75 | 73 | 226
    Ethnicity: Hispanic/Latino | 3 | 5 | 7 | 8 | 23
    Ethnicity: Not Permitted | 0 | 5 | 3 | 3 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 45 | 47 | 45 | 148
  Poland | 0 | 5 | 7 | 5 | 17
  Italy | 0 | 7 | 7 | 4 | 18
  France | 0 | 4 | 1 | 3 | 8
  Germany | 0 | 5 | 4 | 7 | 16
  Spain | 0 | 9 | 13 | 8 | 30
  Russia | 0 | 9 | 7 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The PFS was defined as the time from the date of randomization to the earliest event time of: a) death regardless of cause, or b) first indication of disease progression. PFS was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: Randomization up to 27 months
Population: Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRI + SIM 700 mg (Part A) | FOLFIRI + Placebo (Part B) | FOLFIRI + SIM 200 mg (Part B) | FOLFIRI + SIM 700 mg (Part B)
Number analyzed (Participants) | 11 | 80 | 85 | 84
months | 5.7 [1.8 to 10.0] | 5.8 [4.9 to 9.0] | 5.4 [3.4 to 5.6] | 5.5 [4.0 to 7.1]
Statistical Analysis 1: Comparison: FOLFIRI + Placebo (Part B) vs FOLFIRI + SIM 200 mg (Part B); The null hypothesis was that the hazard ratio (HR) equals to 1 between SIM treatment arm and placebo, while the alternative hypothesis was that HR was less than 1. The HR (95% confidence interval [CI]) and p-value (for comparison between SIM treatment arm and placebo) were based on two-sided log-rank test, stratified based on the 2-level Eastern Cooperative Oncology Group (ECOG) performance status (0 or > 0) at randomization; Test type: Superiority; p = 0.0395, Log Rank; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [1.01 to 2.06]
Statistical Analysis 2: Comparison: FOLFIRI + Placebo (Part B) vs FOLFIRI + SIM 700 mg (Part B); The null hypothesis was that the HR equals to 1 between SIM treatment arm and placebo, while the alternative hypothesis was that HR was less than 1. The HR (95% CI) and p-value (for comparison between SIM treatment arm and placebo) were based on two-sided log-rank test, stratified based on the 2-level ECOG performance status (0 or > 0) at randomization; Test type: Superiority; p = 0.1042, Log Rank; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.92 to 1.89]

2. Secondary Outcome: Overall Survival (OS)
Description: The OS is measured as time from date of randomization to death regardless of cause. The OS was analyzed using KM estimates.
Time Frame: Randomization up to 33 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRI + SIM 700 mg (Part A) | FOLFIRI + Placebo (Part B) | FOLFIRI + SIM 200 mg (Part B) | FOLFIRI + SIM 700 mg (Part B)
Number analyzed (Participants) | 11 | 80 | 85 | 84
months | 9.8 [3.5 to 22.3] | 16.3 [12.0 to 19.5] | 10.5 [9.2 to 12.6] | 11.4 [9.7 to 15.6]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response was assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.1) as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD). The ORR was defined as the percentage of participants who achieved a CR or PR.
Time Frame: Randomization up to 27 months
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRI + SIM 700 mg (Part A) | FOLFIRI + Placebo (Part B) | FOLFIRI + SIM 200 mg (Part B) | FOLFIRI + SIM 700 mg (Part B)
Number analyzed (Participants) | 11 | 80 | 85 | 84
percentage of participants | 9.1 [0.2 to 41.3] | 10.0 [4.4 to 18.8] | 5.9 [1.9 to 13.2] | 11.9 [5.9 to 20.8]

ADVERSE EVENTS:
Time Frame: Randomization up to 33 months
Description: Safety Analysis Set included all participants in the Full Analysis Set grouped for analyses with treatment assignments designated according to the actual study drug received.
Arm/Group | FOLFIRI + SIM 700 mg (Part A) | FOLFIRI + Placebo (Part B) | FOLFIRI + SIM 200 mg (Part B) | FOLFIRI + SIM 700 mg (Part B)
Serious Adverse Events (participants affected / at risk) | 4/11 | 27/80 | 24/85 | 17/84
Other Adverse Events (participants affected / at risk) | 11/11 | 76/80 | 80/85 | 79/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI + SIM 700 mg (Part A) (N=11) | FOLFIRI + Placebo (Part B) (N=80) | FOLFIRI + SIM 200 mg (Part B) (N=85) | FOLFIRI + SIM 700 mg (Part B) (N=84)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2 | 2
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Superior vena cava occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI + SIM 700 mg (Part A) (N=11) | FOLFIRI + Placebo (Part B) (N=80) | FOLFIRI + SIM 200 mg (Part B) (N=85) | FOLFIRI + SIM 700 mg (Part B) (N=84)
Anaemia (Blood and lymphatic system disorders) | 3 | 19 | 23 | 18
Leukopenia (Blood and lymphatic system disorders) | 1 | 9 | 13 | 13
Neutropenia (Blood and lymphatic system disorders) | 6 | 35 | 42 | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6 | 10 | 11
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 18 | 16 | 22
Abdominal pain lower (Gastrointestinal disorders) | 0 | 5 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 6 | 8 | 6
Constipation (Gastrointestinal disorders) | 4 | 17 | 18 | 21
Diarrhoea (Gastrointestinal disorders) | 9 | 43 | 36 | 42
Dry mouth (Gastrointestinal disorders) | 1 | 7 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 7 | 4 | 4
Dysphagia (Gastrointestinal disorders) | 2 | 4 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 3 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 9 | 37 | 38 | 42
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 2 | 3 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 17 | 14 | 9
Vomiting (Gastrointestinal disorders) | 5 | 25 | 21 | 23
Asthenia (General disorders) | 2 | 12 | 13 | 12
Axillary pain (General disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 1 | 0 | 1
Catheter site rash (General disorders) | 1 | 0 | 1 | 0
Chest discomfort (General disorders) | 1 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 3 | 1 | 5
Fatigue (General disorders) | 9 | 34 | 38 | 43
Feeling abnormal (General disorders) | 1 | 0 | 1 | 0
Feeling jittery (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 1 | 5
Mucosal inflammation (General disorders) | 3 | 10 | 14 | 7
Oedema peripheral (General disorders) | 0 | 4 | 14 | 10
Pyrexia (General disorders) | 1 | 11 | 10 | 11
Infection (Infections and infestations) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 2
Pneumonia (Infections and infestations) | 1 | 2 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 6 | 5 | 9
Alanine aminotransferase increased (Investigations) | 0 | 4 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 6 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 6 | 4 | 4
International normalised ratio increased (Investigations) | 1 | 2 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 5 | 3 | 3
Weight decreased (Investigations) | 1 | 7 | 9 | 6
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 22 | 14 | 21
Dehydration (Metabolism and nutrition disorders) | 3 | 4 | 5 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 4 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 8 | 8 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 9 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 6
Dizziness (Nervous system disorders) | 1 | 7 | 9 | 13
Dizziness postural (Nervous system disorders) | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 6 | 6 | 8
Headache (Nervous system disorders) | 1 | 4 | 3 | 6
Neuropathy peripheral (Nervous system disorders) | 2 | 5 | 7 | 7
Parosmia (Nervous system disorders) | 1 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 4 | 2 | 3
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 5 | 5 | 4
Depression (Psychiatric disorders) | 1 | 2 | 3 | 3
Insomnia (Psychiatric disorders) | 5 | 9 | 5 | 8
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 5 | 3 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 10 | 10 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 9 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 5 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 4
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 21 | 20 | 22
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 5 | 2 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2
Skin wrinkling (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Flushing (Vascular disorders) | 2 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 3 | 2 | 4
Peripheral coldness (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years